CLINICAL TRIAL: NCT00354679
Title: Phase II Trial of Irinotecan, Cisplatin, Bevacizumab and Concurrent Radiotherapy in Locally Advanced Esophageal Adenocarcinoma
Brief Title: Irinotecan, Cisplatin, Bevacizumab, Radiation Therapy, and Surgery in Treating Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-013; P30CA008748 (NIH); MSKCC-06013
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; stage III esophageal cancer; stage II esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Bevacizumab; Cisplatin; Irinotecan; Mass Spectrometry; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

ARMS (1):
- Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger (Experimental): Induction therapy: Patients receive cisplatin IV over 30 minutes and irinotecan hydrochloride IV over 30 minutes on days 1, 8, 22, and 29. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 22.
  Combination therapy and radiotherapy: Patients receive cisplatin and irinotecan hydrochloride as in induction chemotherapy on days 43, 50, 64, and 71. Patients also receive bevacizumab IV over 30-90 minutes on days 43 and 64. Patients undergo external beam radiotherapy 5 days a week for 6 weeks beginning on day 43. Surgery: Patients undergo surgery 6-8 weeks after finishing combination therapy and radiotherapy.
  Maintenance therapy: Approximately 6 weeks after surgery, patients receive bevacizumab IV over 30-90 minutes every 3 weeks for 6 months
  Interventions: Biological: bevacizumab; Drug: cisplatin; Drug: irinotecan hydrochloride; Genetic: proteomic profiling; Other: diagnostic laboratory biomarker analysis; Other: mass spectrometry; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: cisplatin
Drug: irinotecan hydrochloride
Genetic: proteomic profiling
Other: diagnostic laboratory biomarker analysis
Other: mass spectrometry
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of esophageal cancer by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and monoclonal antibody therapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bevacizumab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving irinotecan, cisplatin, and bevacizumab together with radiation therapy followed by surgery and bevacizumab works in treating patients with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the toxicity and safety of bevacizumab when given together with cisplatin, irinotecan hydrochloride, and radiotherapy followed by surgery and adjuvant bevacizumab in patients with locally advanced esophageal adenocarcinoma.

Secondary

* Observe the rate of pathologic complete response in patients treated with this regimen.
* Observe overall survival, disease-free survival, and patterns of failure in these patients.
* Clarify toxicity and tolerability of this regimen.
* Evaluate pre-treatment levels of vascular endothelial growth factor in patient serum as a corollary of response to this regimen.
* Correlate serum proteomics data with complete pathologic response.

OUTLINE: This is a nonrandomized, open-label study.

* Induction therapy: Patients receive cisplatin IV over 30 minutes and irinotecan hydrochloride IV over 30 minutes on days 1, 8, 22, and 29. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 22.
* Combination therapy and radiotherapy: Patients receive cisplatin and irinotecan hydrochloride as in induction chemotherapy on days 43, 50, 64, and 71. Patients also receive bevacizumab IV over 30-90 minutes on days 43 and 64. Patients undergo external beam radiotherapy 5 days a week for 6 weeks beginning on day 43.
* Surgery: Patients undergo surgery 6-8 weeks after finishing combination therapy and radiotherapy.
* Maintenance therapy: Approximately 6 weeks after surgery, patients receive bevacizumab IV over 30-90 minutes every 3 weeks for 6 months.

Blood samples are obtained at baseline, after finishing chemoradiotherapy, and prior to maintenance therapy and are examined by the matrix-assisted laser-desorption ionization time of flight (MALDI-TOF) mass spectometry for proteomic profiling.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * T1, N1, M0 or T2-4, any N, M0 esophageal carcinoma that is surgically resectable
  * Disease must be clinically limited to the esophagus or gastroesophageal junction

    * If tumor extends below the gastroesophageal junction into the proximal stomach, 50% of the tumor must involve the distal esophagus or gastroesophageal junction
* No carcinoma in situ (Tis) or tumors determined to be T1, N0 after endoscopy, endoscopic ultrasound, or CT scan
* No gastric cancers with minor involvement of the gastroesophageal junction or distal esophagus
* No metastatic disease, including any of the following:

  * M1a celiac or supraclavicular disease
  * Positive malignant cytology of the pleura, pericardium, or peritoneum
  * Radiographic evidence of distant organ involvement, including lung, liver, bone, or brain
  * No involvement of nonregional lymph nodes including supraclavicular or celiac lymph node metastases that cannot be contained within a radiation field
* No biopsy-proven tumor invasion of the tracheobronchial tree or presence of tracheoesophageal fistula
* No recurrent laryngeal nerve or phrenic nerve paralysis
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* INR ≤ 1.5 (except for patients requiring full-dose warfarin while on bevacizumab)
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT < 2.5 times normal
* Urine protein ≤ 1+ by urinalysis OR < 1 g of protein by 24-hour urine collection
* Calcium < 12 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy (except for basal cell or squamous cell carcinoma of the skin, in situ cervical carcinoma, or superficial transitional cell bladder carcinoma) diagnosed and/or treated within the past 3 years
* No known Gilbert's disease
* No clinically significant hearing loss
* No known hypersensitivity to bevacizumab or other study drugs
* No severe comorbid conditions, including any of the following:

  * Severe uncontrolled diabetes
  * Prior stroke or cerebrovascular disease
  * Uncontrolled infection
  * Nonmalignant illness that precludes study treatment
* No history of serious systemic disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled hypertension (i.e., blood pressure > 160/110 mm Hg on medication)
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
  * Peripheral vascular disease ≥ grade 2
* No significant traumatic injury within the past 28 days
* No evidence of bleeding diathesis or coagulopathy
* No other concurrent medical or psychiatric condition or disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy
* Recovered from prior oncologic or other major surgery
* No major surgery or open biopsy within the past 28 days
* No fine-needle aspiration or core biopsies within the past 7 days
* At least 1 week since prior and no concurrent participation in another experimental drug study (unless Genentech sponsored)
* No other concurrent major surgery
* No other concurrent chemotherapy
* No concurrent sargramostim (GM-CSF)
* No concurrent phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital, Hypericum perforatum (St. John's wort), or other antiepileptic medication

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger: Irinotecan, Cisplatin, Bevacizumab and Concurrent Radiotherapy in Locally Advanced Esophageal Adenocarcinoma
Period: Overall Study
Arm/Group | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger
Started | 34
Completed | 33
Not Completed | 1
Not completed — Patient Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety and Toxicity
Description: All toxicity will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria v3.0.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger
Number analyzed (Participants) | 33
participants
  Anorexia | 1
  Atrial flutter | 1
  CNS cerebrovascular ischemia | 1
  Death not associated with CTCAE term- Death NOS | 1
  Dehydration | 5
  Esophagitis | 7
  Febrile neutropenia | 3
  Hemoglobin | 1
  Hemorrhage, CNS | 1
  Infection, other | 2
  Leukocytes (total WBC) | 2
  Nausea | 2
  Neutrophils/granulocytes (ANC/AGC) | 1
  Pain - Chest wall | 1
  Pain - Extremity-limb | 1
  Perforation, GI- Jejunum | 1
  Phosphate, low (hypophosphatemia) | 1
  Platelets | 1
  Potassium, low (hypokalemia) | 2
  Thrombosis/embolism (vascular access-related) | 1
  Thrombosis/thrombus/embolism | 4
  Vomiting | 2

ADVERSE EVENTS:
Arm/Group | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger
Serious Adverse Events (participants affected / at risk) | 16/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger (N=33)
Anorexia (General disorders) | 1
Atrial flutter (Cardiac disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Ischemia cerebrovascular (Cardiac disorders) | 1
Death not associated with CTCAE term- Death NOS (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 5
Esophagitis (Gastrointestinal disorders) | 7
Febrile neutropenia (General disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
Infection, other (Infections and infestations) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1
Pain - Chest wall (General disorders) | 1
Pain - Extremity-limb (General disorders) | 1
Perforation, GI- Jejunum (Gastrointestinal disorders) | 1
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1
Thrombosis/embolism (vascular access-related) (Cardiac disorders) | 1
Thrombosis/thrombus/embolism (Cardiac disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan, Cisplatin, Bevacizumab, Radiotherapy, & Surger (N=33)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
ALT, SGPT (Blood and lymphatic system disorders) | 9
AST, SGOT (Blood and lymphatic system disorders) | 7
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 8
Constipation (Gastrointestinal disorders) | 4
Creatinine (Metabolism and nutrition disorders) | 2
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dysphagia (Difficulty swallowing) (General disorders) | 2
Esophagitis (Gastrointestinal disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9
Febrile neutropenia (General disorders) | 2
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 21
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 4
Hair loss/alopecia (scalp or body) (General disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 28
Prothrombin time international normalized ratio (Blood and lymphatic system disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 26
Lymphopenia (Blood and lymphatic system disorders) | 31
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 22
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 23
Platelets (Blood and lymphatic system disorders) | 8
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 5
Partial thromboplastin time (Blood and lymphatic system disorders) | 5
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3
Trglycrde, high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2
Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes